CLINICAL TRIAL: NCT05326425
Title: Lazertinib in Patients With Epidermal Growth Factor Receptor Sensitizing Mutation Positive, Metastatic Non-Small Cell Lung Cancer With Asymptomatic or Mild Symptomatic Brain Metastases After Failure of EGFR Tyrosine Kinase Inhibitor
Brief Title: Lazertinib in Patients With NSCLC With Asymptomatic or Mild Symptomatic Brain Metastases After Failure of EGFR TKI.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jin Hyoung Kang (Other)
Responsible Party: Sponsor-Investigator, Jin Hyoung Kang, professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LU20-15
Record Dates: First submitted 2022-03-11; First posted 2022-04-13 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Lung Neoplasms
Keywords: NSCLC; Brain Metastases; Failure of EGFR TKI
MeSH Terms: conditions — Lung Neoplasms; Brain Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- lazertinib(YH25448) (Experimental): lazertinib 240mg, once a day, oral, before disease progression
  Interventions: Drug: lazertinib(YH25448)

INTERVENTIONS:
Drug: lazertinib(YH25448) — - lazertinib 240mg(3tablets, 80mg/1tablet), once a day, oral, before disease progression

SUMMARY:
This is an open-label, single-intervention, multicenter clinical trial in patients with non-small cell lung cancer with asymptomatic or mildly symptomatic brain metastases after failure of EGFR TKI treatment. The objective of this study is as follows.

* Primary objective : intracranial objective response rate (iORR) with RECIST 1.1
* Secondary objectives : intracranial progression free survival(iPFS), Intracranial objective response rate in T790M negative, isolated CNS progression patient group, overall Objective Rsponse Rate(ORR), duration of response(DoR), disease control rate(DCR), treatment failure pattern): intracranial progression or extracranial progression or both, salvage intracranial treatment rate, safety and tolerability

DETAILED DESCRIPTION:
Patients who eligible the inclusion/exclusion criteria should take lazertinib 240 mg (80 mg, 3 tablets) once a day at the same time as possible on an empty stomach before meals. One cycle of treatment is defined as 42 days of continuous administration, and the tumor response by RECIST 1.1 will be evaluated every 1 cycle for the 1st, 2nd, 3rd, and 4th evaluation, and every 2 cycles from the 5th evaluation thereafter. .

If the investigator decides to reduce the dose due to an adverse drug reaction during the administration of lazertinib 240 mg, the dose may be reduced to 160 mg (80 mg, 2 tablets) of lazertinib.

Efficacy and safety will be evaluated by administering lazertinib 240 mg to patients with measurable brain metastasis or newly confirmed metastatic non-small cell lung cancer after failure of treatment with gefitinib, erlotinib, or afatinib after EGFR mutation is confirmed.

ELIGIBILITY:
Inclusion Criteria

* Patients who voluntarily provided written informed consent prior to participation in the clinical trial and genetics and/or exploratory studies
* Male or female, 20 years of age or older(Female patients must agree to the use of appropriate contraceptive methods and not be lactating, and for women of childbearing age, there must be evidence that the pregnancy test is negative prior to initiation of dosing)
* Histologically or cytologically confirmed locally advanced or metastatic non-small cell lung cancer patients. This may occur as systemic recurrence after prior surgery for early stage disease or patients may be newly diagnosed with stage IIIB/C or IV disease.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-2, with no deterioration in the last 2 weeks
* Life expectancy judged by the Investigator of at least 3 months
* Asymptomatic or mild symptomatic brain metastases progressed or newly confirmed patients
* For one or more intracranial measurable disease, the maximum baseline diameter is measured to be 10mm or more on CT or MRI, and this lesions can be ccurately measured. (The target lesion that has received previous local therapy should not be considered as measurable. However, new CNS lesion after more than 3 months of previous local therapy could be considered as target lesion. )
* Confirmed sensitizing EGFR mutation prior to administration of gefitinib, erlotinib, or afatinib (L858R, Exon 19 deletion, G719X and L861Q mutations chould be confirmed as a record)
* Failure after one regimen of EGFR TKI treatment. Past treatment history for locally advanced or metastatic NSCLC limited to one regimen of EGFR TKI treatment (gefitinib, erlotinib, or afatinib) and/or one palliative cytotoxic chemotherapy regimen.
* Those who have been confirmed status of T790M mutations in tissues or blood after EGFR TKI failure (T790M positive or negative should be confirmed as a record)

Exclusion Criteria

* Prior treatment with lazertinib
* Prior treatment with investigational drugs in other clinical trials within 30 days prior to the first administration
* Patients who received cytotoxic chemotherapy for the treatment of advanced non-small cell lung cancer or other anticancer drugs other than EGFR TKI within 14 days prior to the first administration of the investigational drug
* Prior local-regional therapy within 4 weeks prior to Day 1 of trial treatment (e.g., major surgery, radiation therapy [with the exception of palliative bone-directed radiotherapy and radiotherapy administered to superficial lesions], hepatic arterial embolization, transcatheter arterial chemoembolization, chemoembolization, radiofrequency ablation, percutaneous ethanol injection, or cryoablation)
* Patients currently receiving drugs or herbal supplements known as inhibitors or inducers of CYP3A4 or who cannot discontinue use at least 1 week prior to the first dose of lazertinib.
* Previous anticancer treatment-related toxicities not recovered to baseline or Grade 0-1 (except alopecia)
* Symptomatic spinal cord compression (However, registration is allowed if steroid treatment is not required within at least 2 weeks before the start of administration of the investigational drug)
* Symptomatic and unstable central nervous system (CNS) or brain metastasis requiring local treatment at screening. (Asymptomatic or mild symptomatic leptomeningeal metastasis is also permitted to be registered)
* Symptomatic or intracranial bleeding that needs treatment
* History of interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD
* Carcinoma other than non-small cell lung cancer, if the investigator is judged to be inadequate to participate in this clinical trial due to evidence of severe or uncontrolled systemic disease, uncontrolled hypertension, or active bleeding tendency, or that it is difficult to follow this protocol. (Screening for chronic disease is not required)
* Any of the following cardiovascular diaseases: A history of congestive heart failure (CHF) of grade 3 or higher according to the New York Heart Association Classification (NYHA) or cardiac arrhythmia requiring treatment/A History of unstable angina or myocardial infarction experienced within 6 months before the first administration of the investigational drug/Left ventricular ejection fraction <50% on recent echocardiography or MUGA scan
* Known human immunodeficiency virus (HIV) infection
* Patient has known active hepatitis B virus(HBV) or hepatitis C virus (HCV) infection
* Patients with refractory nausea and vomiting, chronic gastrointestinal disorders, inability to swallow the product, or undergoing enterectomy deemed to interfere with the proper absorption of lazertinib.
* History of hypersensitivity to drugs
* Clinically significant chronic infection or major medical or mental illness
* Subjects with any concurrent medical condition or disease that will potentially compromise the conduct of the study at the discretion of the Investigators
* History of allogeneic hematopoietic stem cell transplantation, history of whole blood transfusions that did not remove leukocytes within 120 days before the date of collection of genetics specimens

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-06-23 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Intracranial objective response rates (iORR) (RECIST1.1) | From date of the first administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  iORR will be evaluated according to RECIST v1.1 after IP administration and Response data will be used for the primary endpoint.

SECONDARY OUTCOMES:
intracranial progression free survival, iPFS | Up to 2 years
  the date of onset of objective intracranial disease progression or death of any cause, whichever occurs first.
iORR in T790M negative, isolated CNS progression patient group | From date of the first administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  iORR will be evaluated according to RECIST v1.1 after IP administration
overall ORR | From date of the first administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  ORR will be evaluated according to RECIST v1.1 after IP administration.
duration of response, DoR | Up to 2 years
  Duration from the date of the first documented confirmatory response(CR or PR) to the date of documented disease progression or death (equivalent to the date of the PFS event)
disease control rate, DCR | Up to 2 years
  the percentage of subjects whose response is CR, PR, responding, or SD.
overall survival, OS | Up to 2 years
  the period from the first administration of the investigational drug to the date of death from any cause.
treatment failure pattern | From date of the first administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  intracranial progression or extracranial progression or both
salvage intracranial treatment rate | Up to 2 years
  the percentag of subjects who received salvage treatment(surgery or radiation therapy) due to intracranial disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Hyoung Kang, Study Chair — Seoul St. Mary's Hospital, The Catholic University of Korea
Locations (6):
- South Korea (6):
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul St. Mary's Hospital, Catholic University of Korea, Seoul
  - Yonsei University Health System, Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Goss G, Tsai CM, Shepherd FA, Ahn MJ, Bazhenova L, Crino L, de Marinis F, Felip E, Morabito A, Hodge R, Cantarini M, Johnson M, Mitsudomi T, Janne PA, Yang JC. CNS response to osimertinib in patients with T790M-positive advanced NSCLC: pooled data from two phase II trials. Ann Oncol. 2018 Mar 1;29(3):687-693. doi: 10.1093/annonc/mdx820. PMID 29293889
- [Result] Yun J, Hong MH, Kim SY, Park CW, Kim S, Yun MR, Kang HN, Pyo KH, Lee SS, Koh JS, Song HJ, Kim DK, Lee YS, Oh SW, Choi S, Kim HR, Cho BC. YH25448, an Irreversible EGFR-TKI with Potent Intracranial Activity in EGFR Mutant Non-Small Cell Lung Cancer. Clin Cancer Res. 2019 Apr 15;25(8):2575-2587. doi: 10.1158/1078-0432.CCR-18-2906. Epub 2019 Jan 22. PMID 30670498
- [Result] Ahn MJ, Han JY, Lee KH, Kim SW, Kim DW, Lee YG, Cho EK, Kim JH, Lee GW, Lee JS, Min YJ, Kim JS, Lee SS, Kim HR, Hong MH, Ahn JS, Sun JM, Kim HT, Lee DH, Kim S, Cho BC. Lazertinib in patients with EGFR mutation-positive advanced non-small-cell lung cancer: results from the dose escalation and dose expansion parts of a first-in-human, open-label, multicentre, phase 1-2 study. Lancet Oncol. 2019 Dec;20(12):1681-1690. doi: 10.1016/S1470-2045(19)30504-2. Epub 2019 Oct 3. PMID 31587882
- [Derived] Hong MH, Choi YJ, Ahn HK, Lim SM, Keam B, Kim DW, Kim TM, Youk J, Kim YJ, Hwang S, Kim S, Kim JW, Kim HR, Kang JH. Lazertinib in EGFR-Variant Non-Small Cell Lung Cancer With CNS Failure to Prior EGFR Tyrosine Kinase Inhibitors: A Nonrandomized Controlled Trial. JAMA Oncol. 2024 Oct 1;10(10):1342-1351. doi: 10.1001/jamaoncol.2024.2640. PMID 39145962